CLINICAL TRIAL: NCT05998265
Title: A Randomised, Controlled, Open-Label, Multi-Centre Study to Evaluate the Efficacy of FeetMe® Home-Bases Rehabilitation Program in Comparison to Conventional Physiotherapy in Patients With Parkinson's Disease Using Connected Insoles
Acronym: Re-Connect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: FeetMe (Industry)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A00150-45
Record Dates: First submitted 2023-08-03; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
Keywords: Rehabilitation; Remote monitoring; Physical therapy; Connected insoles
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- FeetMe Rehabilitation arm (Experimental)
  Interventions: Device: FeetMe rehabilitation
- Conventional physiotherapy arm (Active Comparator)
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Device: FeetMe rehabilitation — Home based rehabilitation program with real time biofeedback using a connected device
  Arms: FeetMe Rehabilitation arm
Other: Physiotherapy — Conventional physiotherapy as prescribed by the neurologists
  Arms: Conventional physiotherapy arm

SUMMARY:
The goal of this clinical trial is to compare home based rehalitation program with real time biofeeback versus conventional physiotherapy on the gait velocity in Parkinson disease. The main question[s] it aims to answer are:

• How do the interventions afftect the gait velocity of the participants at week 12 ? Participants will be randomized to either follow prescribtional physiotherapy or FeetMe rehabilitation programs during the first 12 weeks.

At the end of 12 weeks, participants will choose in which arm they want to pursue for 12 aditionnal weeks.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study.
* Male or female patients between 40 to 70 years of age, inclusive.
* Body weight range of 40 kg to120 kg and a body mass index (BMI) of 18 to 34 kg/m2.
* Diagnosis of Idiopathic Parkinson's disease (PD) according to UK Brain Bank Criteria (2/3 symptoms), with Hoehn and Yahr (H&Y) staging level 2, 2.5 or 3.
* Disease onset of at least 3 years prior to enrolment.
* Patients with a history of 50% of levodopa responsiveness based on motor signs.
* On stable treatment of PD medication for at least 30 days before screening and with no expected major changes during the first 3 months of the study.
* Prescription for physiotherapy available.
* Ability to walk without aid for at least 6 minutes.
* Shoe size between 35 - 46 (European Standard).
* Intact skin on feet.
* Adequate visual and auditory acuity to perform the rehabilitation program and the assessments in the Investigator's judgement.
* Comfortable with the use of a smartphone. If assistance is required for the use of FeetMe technology, a caregiver or volunteer is fully available to assist the patient.
* Willingness to be regularly contacted via phone-calls.
* Willingness to suspend conventional physiotherapy treatment and start the FeetMe rehabilitation program, if applicable.
* French speaker.

Exclusion Criteria:

* Medical history indicating a Parkinsonian syndrome other than idiopathic PD.
* Unable to walk without walking aid or presence of an injury preventing the patient to walk.
* Any relevant comorbidity or vestibular/visual dysfunctions limiting locomotion or balance.
* Clinically significant comorbidities which in the judgement of the investigator may preclude the reliable gait assessment of the patient.
* Patients with poor wound healing or broken skin on the feet.
* Patients with foot implants.
* Montreal Cognitive Assessment (MoCA) score ≤ 24/30.
* Patients with dementia.
* Patients with apathy.
* Participation in another clinical trial with an investigational drug/ therapeutic within the three months before screening and during the study, unless agreed by the Sponsor.
* Patients who had Lee Silverman Voice Treatment (LSVT) Big therapy within the past 12 months or have it planned during the course of the study.
* Patients with Deep Brain Stimulation planned during the first 12 weeks of the study.
* Patients with pacemakers.
* Patients performing vigorous exercise > three times a week, 30 mins or more per session.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Gait velocity | Week 12
  Change from baseline to Week 12 (Visit 3) in gait velocity (cm/s) assessed during the 6 Minutes Walk-Test (6MWT).

SECONDARY OUTCOMES:
Stance time variability | Week 12
  Change from baseline to Week 12 (Visit 3) in Stance Time Variability assessed during the 6MWT.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT05998265/Prot_000.pdf
  • Informed Consent Form (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT05998265/ICF_001.pdf